CLINICAL TRIAL: NCT00413387
Title: Double Blind, Double Dummy, Multinational, Multicentre, Parallel-Group Design Clinical Trial of the Efficacy and Tolerability of CHF 1535 (Beclomethasone Dipropionate 100 µg + Formoterol 6 µg) pMDI Via HFA-134a Vs. Budesonide 160 µg + Formoterol 4,5 µg Dry Powder Via Turbuhaler® (Symbicort®) in the 12-Week Treatment of Adult Patients With Moderate to Severe Persistent Asthma
Brief Title: Efficacy and Tolerability of Beclomethasone Dipropionate 100 µg + Formoterol 6 µg pMDI Via HFA-134a Vs. Budesonide 160 µg + Formoterol 4,5 µg Dry Powder Via Turbuhaler®. (Symbicort®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Gabriele Nicolini, Chiesi Farmaceutici
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC/PR/033011/002/03
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Combinations; Inhaled therapy; Corticosteroids; Long acting bronchodilators; Beclomethasone; Formoterol; Budesonide
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): chf1535
  Interventions: Drug: beclomethasone dipropionate plus formoterol fumarate combination
- 2 (Active Comparator): Symbicort
  Interventions: Drug: budesonide plus formoterol combination

INTERVENTIONS:
Drug: beclomethasone dipropionate plus formoterol fumarate combination — 100mcg beclomethasone diproprionate plus 6 mcg formoterol
  Arms: 1
Drug: budesonide plus formoterol combination — 200mcg budesonide plus 6 mcg formoterol
  Arms: 2

SUMMARY:
The aim of this study was to compare the efficacy and tolerability of the fixed combination beclomethasone/formoterol pMDI with that of budesonide/formoterol dry powder via Turbuhaler.

DETAILED DESCRIPTION:
Asthma is a chronic disease that is estimated to affect over 25 million people both in the U.S. and in Europe (i.e. approximately 10% of the total population). Pharmacological therapy is used to treat reversible airway obstruction, inflammation and hyper-reactivity. Medications include preventive treatments in forms of antinflammatory/antiallergic agents (i.e. glucocorticosteroids, leukotriene antagonists, cromolyn sodium) and reliever treatments, in forms of bronchodilators (i.e. β-adrenergic agonists, anticholinergics). In patients treated with inhaled glucocorticosteroids whose asthma is not fully controlled, national and international guidelines recommend a stepwise approach. Recent evidence-based clinical trials show that the addition of a LABA to inhaled glucocorticosteroids is more beneficial in terms of asthma control than increasing the dose of corticosteroids alone.

COMPARISONS: CHF 1535 (BECLOMETHASONE DIPROPIONATE 100 µg+ FORMOTEROL 6 µg) pMDI via HFA-134a compared to SYMBICORT (BUDESONIDE 160 µg + FORMOTEROL 4,5 µg).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe persistent asthma for at least 6 months, according to GINA revised version 2002 guidelines:

  * Forced expiratory volume (FEV1) or peak expiratory flow rate (PEFR) > 50% and < 80% of the predicted normal;
  * Asthma not adequately controlled with the current therapies, defined as presence of daily asthma symptoms > once a week and night-time asthma symptoms > twice a month, and daily use of short-acting β2-agonists. These findings are to be based on recent medical history and are to be confirmed in the 2-week run-in period.

    * Treatment with inhaled corticosteroids at a daily dose ≤ 1000 μg of BDP or equivalent. The daily dose of inhaled corticosteroids taken at visit 1 will be assessed taking into account the following ratios between the doses of the different steroids: fluticasone propionate : BDP CFC = 1 : 2; budesonide : BDP CFC = 4 : 5; flunisolide : BDP CFC = 1 : 1. The ratios between inhaled steroids are irrespective of the formulations (i.e. spray aerosol or powder) used. When BDP is given in the new extra-fine HFA-134a formulation (as QVAR®, 3M Healthcare), the ratio with BDP CFC is set as 2 : 5. Therefore, the maximum allowed daily dose of inhaled corticosteroids at study entry will be: budesonide 800 μg, fluticasone propionate 500 μg, flunisolide 1000 μg, BDP 1000 mcg, BDP HFA extra-fine 400 μg.
    * Positive response to the reversibility test in the screening visit, defined as an increase of at least 12% (or, alternatively, of 200mL) from baseline value in the measurement of FEV1 30 minutes following 2 puffs (2 x 100 µg) of inhaled salbutamol administered via pMDI. The reversibility test can be avoided in patients having a documented positive response in the previous 6 months.
    * A co-operative attitude and ability to be trained to correctly use the metered dose inhalers and to complete the diary cards.
    * Written informed consent obtained.
    * At the end of the 2-week run-in period, the presence of daily asthma symptoms (of at least mild intensity) and nighttime asthma symptom (of at least mild intensity) > once a week, as well as of daily use of relief salbutamol is to be confirmed by reviewing the diary cards for run-in

Exclusion Criteria:

* Inability to carry out pulmonary function testing;

  * Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the National Heart Lung and Blood Institute/World Health Organisation (NHLBI/WHO) Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (30);
  * History of near fatal asthma;
  * Evidence of severe asthma exacerbation or symptomatic infection of the airways in the previous 8 weeks;
  * Three or more courses of oral corticosteroids or hospitalisation due to asthma during the previous 6 months;
  * Patients treated with long-acting β2-agonists, anticholinergics and antihistamines during the previous 2 weeks, with topical or intranasal corticosteroids and leukotriene antagonists during the previous 4 weeks;
  * Patients who have changed their dose of inhaled corticosteroids during the previous 4 weeks, or treatment with inhaled corticosteroids at a daily dose > 1000 μg of BDP or equivalent (except for extra-fine formulations, see inclusion criteria);
  * Current smokers or recent (less than one year) ex-smokers, defined as smoking at least 10 cigarettes/day;
  * History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, cardiac arrhythmias;
  * Diabetes mellitus;
  * Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG) during the previous six months;
  * Patients with an abnormal QTc interval value in the ECG test, defined as > 450 msec in males or > 470 msec in females;
  * Other haemodynamic relevant rhythm disturbances (including atrial flutter or atrial fibrillation with ventricular response, bradycardia (≤ 55 bpm), evidence of atrial-ventricular (AV) block on ECG of more than 1st degree;
  * Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g. active peptic ulcer), neurological or haematological autoimmune diseases;
  * Cancer or any chronic diseases with prognosis < 2 years;
  * Pregnant or lactating females or females at risk of pregnancy, i.e. those not demonstrating adequate contraception (i.e. barrier methods, intrauterine devices, hormonal treatment or sterilization). A pregnancy test is to be carried out in women of a fertile age.
  * History of alcohol or drug abuse;
  * Patients treated with monoamine oxidase inhibitors, tricyclic antidepressants or beta-blockers as regular use;
  * Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
  * Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
  * Patients who received any investigational new drug within the last 12 weeks;
  * Patients who have been previously enrolled in this study;
  * At the end of the run-in period, patients will not be admitted to the treatment period in the case of an increase of PEFR (L/sec) measured at the clinics at the end of the run-in period > 15% in respect of values measured at the start of the run-in period;
  * Patients with asthma exacerbations during the run-in period will also be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2004-09; Primary Completion 2005-08 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Morning Peak Expiratory Flow (PEF) daily measured by patients. | morning approximately 8:00

SECONDARY OUTCOMES:
Evening PEF measured by patients daily. | evening approximately 20:00
FEV1 measured by patients daily. | morning and evening
Standard pulmonary function tests measured at clinics at 2, 4, 8 and 12 weeks. | morning before drug intake
Change in FEV1 and PEF from pre-dose to 5, 15, 30 and 60 minutes after study drug intake at week 0 and 12. | morning post drug intake
Symptoms scores measured by patients daily. | morning and evening
symptoms'free days measured by patients daily. | daily
Use of relief salbutamol measured by patients daily. | daily
Frequency of asthma exacerbations evaluated at 2, 4, 8 and 12 weeks. | morning of the visits retrospective assessment
Adverse event and adverse drug reaction daily. | morning of visits retrospective assesment
ECG (with QTc interval)at 0 and 12 weeks. | morning of start and end of treatment visits
Vital signs (heart rate and blood pressure) at 2, 4, 8 and 12 weeks | morning of visits
Use of relief salbutamol. | daily
Frequency of asthma exacerbations. | at visits

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M. Fabbri, MD, Study Chair — Department of Resipiratory Diseases - University of Modena and Reggio Emilia, Modena, Italy; Maurizio A. Vignola, MD, Study Chair — Institute of Lung Pathophysiology, National Research Council, Palermo, Italy
Locations (13):
- Ambulance For Paediatric and Pulmonology, Vienna, Austria
- Poland (6):
  - Nzoz "Medex"Poradnia Alergologiczna, Bielsko-Biala
  - Centrum Uslug Medycznych, Krakow
  - Centrum Alergologii, Lodz
  - Prywatny Gabinet Lekarski, Lodz
  - Uniwersytet Medyczny, Lodz
  - Nzoz Lekarze Specjalisci, Wroclaw
- Ukraine (6):
  - Internal Medicine Department, Dniepropetrovsk State Medical Academy. City Clinical Hospital no. 4, Dniepropetrovsk
  - Institute of Therapy, Ukranian Academy of Medical Science. Pulmonological Departement, Kharkiv
  - Kharkov Regional Clinical Hospital. Pulmonological and Allergological Department, Kharkiv
  - Institute of Phthisiology and Pulmonology Academy of Medical Science of the Ukraine, Pulmonology Departement, Kiev
  - Institute of Phthisiology and Pulmonology Academy of Medical Science of the Ukraine. Department of Diagnostic, Therapy and Clinical Pharmacology of Lung Diseases, Kiev
  - Kiev Medical Academy of Postdiploma Education. Department of Medical Genetics, Clinical Immunology and Allergology, Kiev

REFERENCES:
- [Result] Papi A, Paggiaro PL, Nicolini G, Vignola AM, Fabbri LM; Inhaled Combination Asthma Treatment versus SYmbicort (ICAT SY) Study Group. Beclomethasone/formoterol versus budesonide/formoterol combination therapy in asthma. Eur Respir J. 2007 Apr;29(4):682-9. doi: 10.1183/09031936.00095906. Epub 2006 Nov 15. PMID 17107988